CLINICAL TRIAL: NCT02182921
Title: Evaluation of Surgical Outcomes of Cataract Surgery
Brief Title: Evaluation of Cataract Surgery Outcome
Status: Recruiting | Type: Observational
Sponsor: Evidence Based Cataract Study Group (Other)
Responsible Party: Principal Investigator, xiangjiazhu, MD, Evidence Based Cataract Study Group
Other Study IDs: NSFC/YOUNG-81100653
Record Dates: First submitted 2014-06-24; First posted 2014-07-08 (Estimated); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Cataract; High Myopia
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to evaluate the visual outcome of the cataract surgery, including best uncorrected and corrected visual acuity, spherical equivalent, wavefront aberration and other measurements.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cataract
* Must be able to cooperate with the ophthalmic examination

Exclusion Criteria:

* Clinical diagnosis of mental illness
* Mentally disabled

Max Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Medical centre: Eye and ENT Hospital of Fudan University
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2013-08; Primary Completion 2026-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in visual acuity at one month after cataract surgery | Follow-up until one month after surgery
Change from baseline in spherical equivalent at one month after cataract surgery | Follow-up until one month after surgery
Change from baseline in visual acuity at six months after cataract surgery | Follow-up until six months after surgery
Change from baseline in spherical equivalent at six months after cataract surgery | Follow-up until six months after cataract surgery

SECONDARY OUTCOMES:
Change from baseline in wavefront aberration at one month after cataract surgery | Follow-up until one month after surgery
Change from baseline in contrast sensitivity at one month after cataract surgery | Follow-up until one month after surgery
Change from baseline in intraocular light scattering at one month after cataract surgery | Follow-up until one month after surgery
Change from baseline in wavefront aberration at six months after cataract surgery | Follow-up until six months after surgery
Change from baseline in contrast sensitivity at six months after cataract surgery | Follow-up until six months after surgery
Change from baseline in intraocular light scattering at six months after cataract surgery | Follow-up until six months after surgery

OTHER OUTCOMES:
The difference between attempted and achieved refractive correction at one month after cataract surgery | Follow-up until one month after surgery
The difference between attempted and achieved refractive correction at six months after cataract surgery | Follow-up until six months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yi Lu, MD, Study Chair — Eye and ENT Hospital of Fudan University; Xiangjia Zhu, MD, Study Director — Eye and ENT Hospital of Fudan University; Jin Yang, MD, Study Director — Eye and ENT Hospital of Fudan University; Keke Zhang, MD, Principal Investigator — Eye and ENT Hospital of Fudan University; Wenwen He, MD, Principal Investigator — Eye and ENT Hospital of Fudan University
Locations (1):
- Eye and ENT Hospital of Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhou J, Chen Y, Meng J, Cheng K, Qi J, Du Y, Yao Y, Lu Y, He W, Zhu X. Comparative analysis of iris blood flow after first-eye and second-eye cataract surgeries: insights into increased pain perception in the second eye. BMJ Open Ophthalmol. 2025 Aug 19;10(1):e002162. doi: 10.1136/bmjophth-2025-002162. PMID 40835236
- [Derived] Chen C, Zhou J, Cheng K, Hu X, Zhu M, Du Y, Meng J, Lu Y, He W, Zhu X. Lens position change following cataract surgery in eyes with thick lenses: an SS-OCT based study. Br J Ophthalmol. 2025 Sep 23;109(10):1120-1125. doi: 10.1136/bjo-2025-327414. PMID 40461064
- [Derived] Yao Y, Meng J, He W, Zhang K, Wei L, Cheng K, Lu Y, Zhu X. Associations between anterior segment parameters and rotational stability of a plate-haptic toric intraocular lens. J Cataract Refract Surg. 2021 Nov 1;47(11):1436-1440. doi: 10.1097/j.jcrs.0000000000000653. PMID 34675151
- [Derived] Lu Q, Wei L, He W, Zhang K, Wang J, Zhang Y, Rong X, Zhao Z, Cai L, He X, Wu J, Ding D, Lu Y, Zhu X. Lens Opacities Classification System III-based artificial intelligence program for automatic cataract grading. J Cataract Refract Surg. 2022 May 1;48(5):528-534. doi: 10.1097/j.jcrs.0000000000000790. PMID 34433780
- [Derived] Zhu X, Lu Q, Yao Y, Xu X, Lu Y. Intraoperative Pain Sensation During Cataract Surgery: Why Does Timing Matter? Curr Eye Res. 2021 Jul;46(7):971-977. doi: 10.1080/02713683.2020.1857776. Epub 2020 Dec 15. PMID 33249933
- [Derived] Lu Q, He W, Lu Y, Zhu X. Morphological features of anterior segment: factors influencing intraocular pressure after cataract surgery in nanophthalmos. Eye Vis (Lond). 2020 Sep 9;7:47. doi: 10.1186/s40662-020-00212-4. eCollection 2020. PMID 32974413
- [Derived] Zhu X, Qi J, He W, Zhang S, Zhang K, Lu Q, Lu Y. Early transient intraocular pressure spike after cataract surgery in highly myopic cataract eyes and associated risk factors. Br J Ophthalmol. 2020 Aug;104(8):1137-1141. doi: 10.1136/bjophthalmol-2019-315117. Epub 2019 Nov 8. PMID 31704699
- [Derived] Zhu X, He W, Zhang K, Lu Y. Factors influencing 1-year rotational stability of AcrySof Toric intraocular lenses. Br J Ophthalmol. 2016 Feb;100(2):263-8. doi: 10.1136/bjophthalmol-2015-306656. Epub 2015 Jun 18. PMID 26089212